CLINICAL TRIAL: NCT05360667
Title: The Clinical Effectiveness of Exergame-based Exercise Training in the Prevention of Fragile Syndrome and Sarcopenia Among Elders in Rural Long-term Care Facilities
Brief Title: Using Exergame-based Program in Elders of Rural LTCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cishan Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Principal Investigator, Sheng-Hui Tuan, Attending physicain, Cishan Hospital, Ministry of Health and Welfare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-01
Record Dates: First submitted 2022-04-24; First posted 2022-05-04 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Sarcopenia; Frailty; Long Term Care Facility
Keywords: long-term care; exergame; RingFit Adventure; elderly; appendicular skeletal muscle index; Study of Osteoporotic Fractures Index
MeSH Terms: conditions — Sarcopenia; Frailty | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: @Intervention group: The program consists of PRT and functional movement of the four extremities but mainly the upper limbs. We used RFA to deliver the program. The exergame-based exercise were performed two times per week, at least 48 h apart from each training session, 50 min per session (10 min each for a warm-up and cool-down and 30 min for the main program), for 12 weeks, and will be supervised by a therapist.
  @Control group: Participants in the control group received standard care that applied as usual in the LTCFs, in the way of group activities, including calisthenics (that could be performed in the sitting position), horticultural therapy, and group static activities (e.g., tabletop games). The programs were performed two times per week for approximately 30-60 min, depending on the activity, and will be led by a therapist.
Who Masked: Outcomes Assessor
Masking Description: Because of the design of the study and the nature of the interventions, blinding the staff and participants of the LTCFs is impossible. The assessors, measuring the outcomes, and the interpreter, analyzing the data, will be blinded in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention in this group is standard care plus plus exergame-based multicomponent training program
  Interventions: Other: Standard care plus plus Exergame-based multicomponent training program
- Control group (Sham Comparator): The control group receives usual care in the LTCFs.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Standard care plus plus Exergame-based multicomponent training program — The program contains PRT and functional movement of the four extremities but mainly upper limbs. We will use the commercialized exergame Ringfit Adventure (RFA) to deliver the program.
  RFA is a ﬁtness action role-playing game. The player advances the story while exercising as the movement of the player is linked to the main character on the screen. The movements of the player and battle actions are based on performing certain physical activities using the Ring-Con and Leg Strap. RFA itself could estimate the optimal exercise intensity for each player and performs ﬁne-tuned up-and downregulation based on these physiological feedbacks. Therefore, it has become possible to provide an appropriate amount of exercise for all generations from children to the elderly.
  The standard care is applied as usual in our LTCF. (descriped as the below in the control group)
  Arms: Intervention group
Other: Standard care — The standard care in the control group is applied as usual in our LTCF, in the way of group activity, including calisthenics (that could be done in sitting position), horticultural therapy, and group activity of peace (like tabletop games). The programs are performed twice per week, about 30 to 60 minutes (depends on different activity), leading by a therapist.
  Arms: Control group

SUMMARY:
Background:

Sarcopenia is the progressive loss of skeletal muscle mass and decline of muscle function associated with aging. Frailty is defined as a clinically recognizable state of increased vulnerability resulting from aging-associated decline in reserve and function across multiple physiologic systems. Resistant, aerobic, and multi-component exercise could improve muscle strength and function in older adults. Some policies have been proposed and implemented to prevent and delay the frailty and disability among elders in long term care policy in Taiwan. However, due to shortage in healthcare provider, long-term exercise program is difficult to provide in long-term care facilities (LTCF) of countryside in Taiwan.

Method:

This will be a prospective randomized controlled trial comparing an exergame-based multicomponent training (Exergame-based REH) to standard of care in older users of LTCF in rural Kaohsiung city, Taiwan. Participants in the intervention group will receive Exergame-based REH for 12 weeks, while participants in the control group will receive standard care that routinely applied in the LTFC as usual. The Exergame-based REH contains progressive resistance training and functional movement of the four extremities but mainly upper limbs. The investigators will use the Ringfit Adventure to deliver the program. The Exergame-based REH will be performed twice per week, at least 48 hours apart from each training session, 50 minutes per time, for a total 12 weeks. Criteria of sarcopenia including (1) handgrip strength of dominant hand, (2) walking speed, and (3) appendicular skeletal muscle mass index of 4 extremities, and Study of osteoporotic fractures index, will be measured as primary outcomes. (1) Range of motions in dominant upper extremity, (2) maximal voluntary isometric contraction of biceps/triceps brachial muscles of dominant side, (3) box and block test, (4) Sonographic thickness of Biceps and Triceps Brachii muscles, (5) Kihon checklist-Taiwan version, (6) 36-Item Short Form Survey questionnaire, and (7) brain health test, will be measured as secondary outcomes before and after the programs.

Anticipated benefits:

The Exergame-based REH could enhance the motivation toward exercise of older adults. It could also increase muscle mass, strength, functional ability of dominant upper extremity, and health-related quality of life.

DETAILED DESCRIPTION:
Background:

Sarcopenia is the progressive loss of skeletal muscle mass and decline of muscle function associated with aging. The prevalence of sarcopenia among people older than 65 years old in Taiwan is over 20%. Sarcopenia is one of the most important causes of functional decline and loss of independence, even mortality in older adults. Frailty is theoretically defined as a clinically recognizable state of increased vulnerability resulting from aging-associated decline in reserve and function across multiple physiologic systems such that the ability to cope with everyday or acute stressors is comprised. Both sarcopenia and frailty are getting more and more concerns in Taiwan, which is now an aged-society. Resistant, aerobic, and multi-component exercise have been proved to improve muscle strength and function in older adults.

The principles of progressive resistance training and multi-component exercise programs include regular, mass-practiced, mild overwhelming engagement. These principles demand devoting time, workforce, and money to achieve. Staffing constraints and resources shortage have made it challenging to promote regular exercise programs in long-term care facilities. Exergames have been defined as any type of video game that requires the movement of the player's entire body, allowing real-time interaction. Exergames breaks down the barriers of repetitive and monotonous physical exercise since they contain attractive and multisensory game environments with an immersive environment in which the interaction takes place through global body movements. Moreover, the gamified approach and immersive scenarios motivate older people to acquire a greater commitment to the practice of physical and rehabilitative exercises. Therefore, by playing exergames, it reduces staff time for intervention, encourages patients to perform relatively high-energy movements, and increase participants' motivation.

Therefore, investigators in this study aim to evaluate the feasibility and clinical application of a novel exergame-based multicomponent training via Nintendo Switch® Ringfit Adventure (RFA), (which could deliver optimal exercise intensity for each player and perform fine-tuned up- and downregulation based on performance after each game), among older adults in rural care facilities in this current study.

Methods:

The investigators will conduct a prospective randomized controlled trial (RCT) comparing an exergame-based multicomponent training (Exergame-based REH) to standard of care in older users of LTCF in Ci-Shan and Mei-Nong district, Kaohsiung city, Taiwan. Participants in the intervention group will receive standard care with additional exergame-based REH for 12 weeks, while participants in the control group will receive standard care that routinely applied in the long term care facilities as usual. The Exergame-based REH contains progressive resistance training and functional movement of the four extremities but mainly upper limbs. The investigators will use the commercialized exergame Ringfit Adventure (RFA) to deliver the program. The Exergame-based REH will be performed twice per week, at least 48 hours apart from each training session, 50 minutes (10 minutes for warm-up and cool-down, 30 minutes for main program) per time, for a total 12 weeks. Criteria of sarcopenia including (1) handgrip strength of dominant hand (HGS), (2) walking speed, and (3) appendicular skeletal muscle mass index of 4 extremities (ASMMI), and study of osteoporotic fractures index, will be measured as primary outcomes. (1) Range of motions in dominant upper extremity (ROM), (2) maximal voluntary isometric contraction of biceps/triceps brachial muscles of dominant side (MVC of biceps/triceps), (3) box and block test (BBT), (4) Sonographic thickness of Biceps and Triceps Brachii muscles, (5) Kihon checklist-Taiwan version, (6) 36-Item Short Form Survey questionnaire (SF-36), and (7) brain health test (BHT) will be measured as secondary outcomes before, during, and after the programs.

Hypothesis

1. After three months of participating in the Exergame-based REH, the primary outcomes will show statistically significant increase.
2. After three months of participating in the Exergame-based REH, the secondary outcomes will show statistically significant increase.

Flow of the research:

Participants meet the inclusion criteria are first selected from the long term care facilities (including daycare centers and nursing homes) in Chi-Shan and Mei-Nong districts in rural Kaohsiung city.

The participants are classified into the intervention and control group randomly.

All the outcomes measured are done at the baseline (pre-test), 6 weeks after the intervention (mid-term evaluation), and 3 months after the intervention (post-test).

Apparatus in this study:

Nintendo Switch® RingFit Adventrue with RIng-Con and Joy-con. InBody S10 Body Composition & Scale JAMAR Hand Dynamometer MicroFET3 Dynamometer and range of motion evaluator Goniometer Box and Block Test Apparatus A portable LOGIQ e ultrasound (General Electric Company, U.S.A., 2010), equipped with a 5-12 MHz linear array transducer

ELIGIBILITY:
Inclusion Criteria:

* individuals aged ≥60 years
* those living or participating in LTCFs for at least 1 month
* those who can understand and speak Chinese or Taiwanese
* those with sufficient cognitive capacity (judged by the researchers) to give informed consent and participate in the exergame-based REH and data collection
* those who can sit for more than 50 min for training and can complete the measurement of gait speed.

Exclusion Criteria:

* Individuals who have significant cardiopulmonary diseases
* those regularly receiving oxygen supplementation
* those who have uncontrollable hypertension
* those who had a recent infection or fracture or were diagnosed with other diseases that might prohibit them from participating in exercises according to the guidelines of the American College of Sports Medicine.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change of anthropometry and body composition (T2-T0) | Change from baseline appendicular skeletal muscle mass index at the end of the 12th weeks
  We choose bioelectrical impedance analysis to evaluate participants' appendicular skeletal muscle mass. ASMMI was defined as the appendicular skeletal muscle mass (in kilograms) divided by the height squared (in meters squared).
Change of anthropometry and body composition (T1-T0) | Change from baseline appendicular skeletal muscle mass index at the end of the 6th weeks
  We choose bioelectrical impedance analysis to evaluate participants' appendicular skeletal muscle mass. ASMMI was defined as the appendicular skeletal muscle mass (in kilograms) divided by the height squared (in meters squared).
Change of anthropometry and body composition (T2-T1) | Change of appendicular skeletal muscle mass index between the 6th week and the 12th week
  We choose bioelectrical impedance analysis to evaluate participants' appendicular skeletal muscle mass. ASMMI was defined as the appendicular skeletal muscle mass (in kilograms) divided by the height squared (in meters squared).
Dominant Hand Grip Strength (HGS) (T2-T0) | Change from baseline HGS at the end of 12th weeks
  The HGS will be measured by a JAMAR dynamometer (J A Preston, New York, NY) using all five notches. The measurement is done three times and the highest of the three measurements will be recorded. The participants are allowed to rest for 1 min between each measurement.
Dominant Hand Grip Strength (HGS) (T1-T0) | Change from baseline appendicular skeletal muscle mass index at the end of the 6th weeks
  The HGS will be measured by a JAMAR dynamometer (J A Preston, New York, NY) using all five notches. The measurement is done three times and the highest of the three measurements will be recorded. The participants are allowed to rest for 1 min between each measurement.
Dominant Hand Grip Strength (HGS) (T2-T1) | Change of HGS between the end of the 6th week and the 12th week
  The HGS will be measured by a JAMAR dynamometer (J A Preston, New York, NY) using all five notches. The measurement is done three times and the highest of the three measurements will be recorded. The participants are allowed to rest for 1 min between each measurement.
Gait Speed (T2-T0) | Change from baseline gait speed at the end of the 12th weeks
  The participants are asked to walk a 6-m long corridor without a barrier and the usual gait speed calculated by measuring the time spent by a participant as suggested by ASWG.
Gait Speed (T1-T0) | Change from baseline gait speed at the end of the 6th weeks
  The participants are asked to walk a 6-m long corridor without a barrier and the usual gait speed calculated by measuring the time spent by a participant as suggested by ASWG.
Gait Speed (T2-T1) | Change of gait speed between the end of the 6th week and the 12th week
  The participants are asked to walk a 6-m long corridor without a barrier and the usual gait speed calculated by measuring the time spent by a participant as suggested by ASWG.
Study of Osteoporotic Fractures Index (SOF index) (T2-T0) | Change from baseline SOF index at the end of the 12th weeks
  SOF index composes of the following three components: (a) a weight loss of ≥5% during the preceding year (regardless of any intention to lose weight), (b) an inability to rise from a chair five times without using the arms, and (c) an answer of 'no' to the question 'Do you feel full of energy?'. Participants are identified to be frail by the presence of two or more of the components, those with one disability are considered to be in pre-frailty status, and those with none of the above impairments are considered to be robust.
Study of Osteoporotic Fractures Index (SOF index) (T1-T0) | Change from baseline SOF index at the end of the 6th weeks
  SOF index composes of the following three components: (a) a weight loss of ≥5% during the preceding year (regardless of any intention to lose weight), (b) an inability to rise from a chair five times without using the arms, and (c) an answer of 'no' to the question 'Do you feel full of energy?'. Participants are identified to be frail by the presence of two or more of the components, those with one disability are considered to be in pre-frailty status, and those with none of the above impairments are considered to be robust.
Study of Osteoporotic Fractures Index (SOF index) (T2-T1) | Change of SOF index between the end of the 6th week and the 12th week
  SOF index composes of the following three components: (a) a weight loss of ≥5% during the preceding year (regardless of any intention to lose weight), (b) an inability to rise from a chair five times without using the arms, and (c) an answer of 'no' to the question 'Do you feel full of energy?'. Participants are identified to be frail by the presence of two or more of the components, those with one disability are considered to be in pre-frailty status, and those with none of the above impairments are considered to be robust.

SECONDARY OUTCOMES:
Box and Block Test (BBT) | baseline (before intervention), during-test (at the end of 6th week), post-test (at the end of 12th week)
  BBT can be used to measure the unilateral gross manual dexterity in various populations with high test-retest reliability and validity. The setup of BBT comprised a wooden box, divided into two compartments, with 100 wooden blocks inside one compartment.
Biceps and Triceps Brachii Muscle Strength of the dominant side | baseline (before intervention), during-test (at the end of 6th week), post-test (at the end of 12th week)
  We will use the microFET® 3 (Hoggan Health Industries, West Jordan, UT) to The test will bmeasure the maximal voluntary isometric contraction (MVIC) of the biceps and triceps brachii of the dominant side. MicroFET® 3 is an electronic handheld dynamometer that can detect 0-150 lb of force with high reliability and validity(61). The participants lie on the treatment table with their elbows forming a 90° angle to the horizontal such that the arm is perpendicular to the limb. The test will be done under standard positions.
Sonographic thickness of Biceps and Triceps Brachii muscles | baseline (before intervention), during-test (at the end of 6th week), post-test (at the end of 12th week)
  An experienced single operator who is not involved in any further data analysis and is blinded to clinical symptoms, will use a portable LOGIQ e ultrasound (General Electric Company, U.S.A., 2010), equipped with a 5-12 MHz linear array transducer, to measure the muscle thickness under sonography. All the measurements will be done under standard positions.
Measurement of the range of motion (ROM) of the Joints of Dominant Upper Extremity | baseline (before intervention), during-test (at the end of 6th week), post-test (at the end of 12th week)
  The ROMs, including shoulder flexion, abduction, and external rotation; elbow flexion and extension; forearm supination and pronation and wrist flexion and extension, of the dominant upper extremity of the participants are measured. The ROMs measurement is done by a goniometer under standard positions.
General function | baseline (before intervention), during-test (at the end of 6th week), post-test (at the end of 12th week)
  We will use Kihon checklist-Taiwan (KC-T) to indicate the ADLs of the participants in this study. KC-T is a self-reported questionnaire, consisting of 25 items divided into 7 sub-categories: general independence, physical strength, nutrition, oral function, level of social activities outside the home, cognitive function, and risk of depression.
Health-related Quality of Life (HQoL) | baseline (before intervention), during-test (at the end of 6th week), post-test (at the end of 12th week)
  We will use the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) to indicate the HQoL in this study, The SF-36 is a self-assessment validated generic health survey containing 36 items, divided into 8 subscales, including physical functioning, role limitation due to physical problems, bodily pain, general health, vitality, social functioning, role limitation due to emotional problems, and mental health.
Cognitive level | baseline (before intervention), during-test (at the end of 6th week), post-test (at the end of 12th week)
  e will use Brain Health Test (BHT)- brief cognitive test (BHT-Cog) to measure the cognitive level of the participants in this study. The BHT, developed by Taiwan Dementia Society, is a simple dementia screening tool with high validity to assist primary care physicians in identifying patients with cognitive impairment among subjects with memory complaints or at a high risk for dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Hui Tuan, M.D., Principal Investigator — Ci-Shan hospital, Ministry of Health and Welfare
Locations (1):
- Cishan Hospital, Ministry of health and welfare, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and analysed during the current study are not publicly available since the study is just under construction. The data will be available from the primary investigator on reasonable request after the publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after the official publication.
Access Criteria: Please e-mail to the primary investigator on reasonable request after the publication.

REFERENCES:
- [Background] Evans WJ. Skeletal muscle loss: cachexia, sarcopenia, and inactivity. Am J Clin Nutr. 2010 Apr;91(4):1123S-1127S. doi: 10.3945/ajcn.2010.28608A. Epub 2010 Feb 17. PMID 20164314
- [Background] Seene T, Kaasik P, Riso EM. Review on aging, unloading and reloading: changes in skeletal muscle quantity and quality. Arch Gerontol Geriatr. 2012 Mar-Apr;54(2):374-80. doi: 10.1016/j.archger.2011.05.002. Epub 2011 May 31. PMID 21632125
- [Background] Chang CF, Yeh YL, Chang HY, Tsai SH, Wang JY. Prevalence and Risk Factors of Sarcopenia among Older Adults Aged >/=65 Years Admitted to Daycare Centers of Taiwan: Using AWGS 2019 Guidelines. Int J Environ Res Public Health. 2021 Aug 5;18(16):8299. doi: 10.3390/ijerph18168299. PMID 34444047
- [Background] Thomas E, Battaglia G, Patti A, Brusa J, Leonardi V, Palma A, Bellafiore M. Physical activity programs for balance and fall prevention in elderly: A systematic review. Medicine (Baltimore). 2019 Jul;98(27):e16218. doi: 10.1097/MD.0000000000016218. PMID 31277132
- [Background] Hsu HC, Chen CF. LTC 2.0: The 2017 reform of home- and community-based long-term care in Taiwan. Health Policy. 2019 Oct;123(10):912-916. doi: 10.1016/j.healthpol.2019.08.004. Epub 2019 Aug 20. PMID 31455563
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Meekes W, Stanmore EK. Motivational Determinants of Exergame Participation for Older People in Assisted Living Facilities: Mixed-Methods Study. J Med Internet Res. 2017 Jul 6;19(7):e238. doi: 10.2196/jmir.6841. PMID 28684385
- [Background] Jahouh M, Gonzalez-Bernal JJ, Gonzalez-Santos J, Fernandez-Lazaro D, Soto-Camara R, Mielgo-Ayuso J. Impact of an Intervention with Wii Video Games on the Autonomy of Activities of Daily Living and Psychological-Cognitive Components in the Institutionalized Elderly. Int J Environ Res Public Health. 2021 Feb 7;18(4):1570. doi: 10.3390/ijerph18041570. PMID 33562249
- [Background] Gunst M, De Meyere I, Willems H, Schoenmakers B. Effect of exergaming on wellbeing of residents in a nursing home: a single blinded intervention study. Aging Clin Exp Res. 2022 Jan;34(1):151-157. doi: 10.1007/s40520-021-01903-1. Epub 2021 Jun 22. PMID 34156650
- [Background] Sato T, Shimizu K, Shiko Y, Kawasaki Y, Orita S, Inage K, Shiga Y, Suzuki M, Sato M, Enomoto K, Takaoka H, Mizuki N, Kim G, Hozumi T, Tsuchiya R, Otagiri T, Mukaihata T, Furuya T, Maki S, Nakamura J, Hagiwara S, Aoki Y, Koda M, Akazawa T, Takahashi H, Takahashi K, Ohtori S, Eguchi Y. Effects of Nintendo Ring Fit Adventure Exergame on Pain and Psychological Factors in Patients with Chronic Low Back Pain. Games Health J. 2021 Jun;10(3):158-164. doi: 10.1089/g4h.2020.0180. Epub 2021 Apr 22. PMID 33891508
- [Background] Chen GB, Lin CW, Huang HY, Wu YJ, Su HT, Sun SF, Tuan SH. Using Virtual Reality-Based Rehabilitation in Sarcopenic Older Adults in Rural Health Care Facilities-A Quasi-Experimental Study. J Aging Phys Act. 2021 Oct 1;29(5):866-877. doi: 10.1123/japa.2020-0222. Epub 2021 Feb 16. PMID 33596540
- [Background] Choi HJ, Ko CY, Chang Y, Kim GS, Choi K, Kim CH. Development and validation of bioimpedance prediction equations for fat-free mass in unilateral male amputees. PeerJ. 2021 Mar 8;9:e10970. doi: 10.7717/peerj.10970. eCollection 2021. PMID 33732549
- [Background] Bobos P, Nazari G, Lu Z, MacDermid JC. Measurement Properties of the Hand Grip Strength Assessment: A Systematic Review With Meta-analysis. Arch Phys Med Rehabil. 2020 Mar;101(3):553-565. doi: 10.1016/j.apmr.2019.10.183. Epub 2019 Nov 13. PMID 31730754
- [Background] Ensrud KE, Ewing SK, Cawthon PM, Fink HA, Taylor BC, Cauley JA, Dam TT, Marshall LM, Orwoll ES, Cummings SR; Osteoporotic Fractures in Men Research Group. A comparison of frailty indexes for the prediction of falls, disability, fractures, and mortality in older men. J Am Geriatr Soc. 2009 Mar;57(3):492-8. doi: 10.1111/j.1532-5415.2009.02137.x. Epub 2009 Feb 22. PMID 19245414
- [Background] Desrosiers J, Bravo G, Hebert R, Dutil E, Mercier L. Validation of the Box and Block Test as a measure of dexterity of elderly people: reliability, validity, and norms studies. Arch Phys Med Rehabil. 1994 Jul;75(7):751-5. PMID 8024419
- [Background] Stark T, Walker B, Phillips JK, Fejer R, Beck R. Hand-held dynamometry correlation with the gold standard isokinetic dynamometry: a systematic review. PM R. 2011 May;3(5):472-9. doi: 10.1016/j.pmrj.2010.10.025. PMID 21570036
- [Derived] Tuan SH, Chang LH, Sun SF, Li CH, Chen GB, Tsai YJ. Assessing the Clinical Effectiveness of an Exergame-Based Exercise Training Program Using Ring Fit Adventure to Prevent and Postpone Frailty and Sarcopenia Among Older Adults in Rural Long-Term Care Facilities: Randomized Controlled Trial. J Med Internet Res. 2024 Jul 18;26:e59468. doi: 10.2196/59468. PMID 39024000
- [Derived] Tuan SH, Chang LH, Sun SF, Lin KL, Tsai YJ. Using exergame-based exercise to prevent and postpone the loss of muscle mass, muscle strength, cognition, and functional performance among elders in rural long-term care facilities: A protocol for a randomized controlled trial. Front Med (Lausanne). 2022 Dec 13;9:1071409. doi: 10.3389/fmed.2022.1071409. eCollection 2022. PMID 36582297